CLINICAL TRIAL: NCT06534255
Title: A Clinical Trial to Evaluate the Safety, Efficacy, and Pharmacokinetics of MegaLT Injection for Treating Refractory Thrombocytopenia Following Radiotherapy, Chemotherapy, or Transplantation.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MegaLT-2024
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2024-12

CONDITIONS: Refractory Thrombocytopenia
Keywords: Refractory thrombocytopenia; Megakaryocyte
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Intervention Model Description: Subjects will receive cell infusions sequentially according to their enrollment order, with three planned dose levels of: 1×10⁶/kg, 5×10⁶/kg, and 1×10⁷/kg.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MegaLT injection (Experimental): Dosage Form: ex vivo three-dimensional induced umbilical cord blood mononuclear cells differentiated megakaryocyte injection (MegaLT injection).
  Administration Route: Intravenous Infusion Regimen: Single or Multiple Infusions
  Interventions: Biological: MegaLT injection

INTERVENTIONS:
Biological: MegaLT injection — Three dose groups were set: 1×10^6/kg, 5×10^6/kg, and 1×10^7/kg. The dose escalation was carried out in ascending order using a "3+3" design. To ensure participant safety, enrollment followed a "1+2" rule. Specifically, the first participant in each dose group received the cell infusion and was observed for 14 days. If no dose-limiting toxicity (DLT) was observed, the remaining two participants could then be enrolled and receive cell therapy at the same dose level.

SUMMARY:
A study to evaluate the safety, efficacy, and pharmacokinetics of MegaLT in treating refractory thrombocytopenia following radiotherapy, chemotherapy, or transplantation.

DETAILED DESCRIPTION:
A single-center, open-label, dose-escalation study to assess the safety, efficacy, and pharmacokinetics of MegaLT for treating refractory thrombocytopenia following radiotherapy, chemotherapy, or transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 4 and 75 years (inclusive) at screening; gender is not restricted;
* Diagnosed with refractory thrombocytopenia following radiotherapy/chemotherapy or transplantation;
* Adequate organ function：Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) < 2.5*upper limit of normal (ULN); Serum creatinine < 1.5* ULN; Total bilirubin level < 1.5* ULN; Coagulation function: International Normalized Ratio (INR) ≤ 1.5* ULN, Activated Partial Thromboplastin Time (APTT) ≤ 1.5*ULN; Hemoglobin ≥ 60 g/L, or hemoglobin maintained at this level after transfusion; Absolute neutrophil count (ANC) ≥ 1.0×10^9/L;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
* Voluntarily participating in the clinical trial, with full understanding of the trial details and having signed the informed consent form.

Exclusion Criteria:

* Patients with any malignant tumor relapse;
* Pregnant or breastfeeding women;
* Life expectancy less than 3 months;
* Severe infections or severe concurrent conditions such as heart, liver, lung, kidney, neurological, or metabolic diseases;
* History of severe thrombotic events or known thrombotic risk factors. Exceptions: Participants for whom the potential benefits of the study, as determined by the investigator, outweigh the potential risks of thromboembolic events;
* Uncontrolled infectious or other serious diseases, including but not limited to infections (e.g., HIV positive), congestive heart failure, unstable angina, arrhythmias, psychiatric disorders, or conditions that limit the ability to meet study requirements or pose unpredictable risks as judged by the primary physician;
* Active hepatitis B or C infection;
* Refractory thrombocytopenia post-transplant with Grade III-IV acute graft-versus-host disease (GVHD) [according to NIH standards] or severe chronic GVHD (NIH 2014 standards);
* History of organ transplantation or planned organ transplantation (excluding hematopoietic stem cell transplantation);
* Participation in another clinical study within 30 days prior to the baseline visit, involving any investigational drug or device; observational studies are allowed;
* Any other conditions deemed by the investigator to make the participant unsuitable for the clinical trial.

Ages: 4 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2026-05-22 (Estimated)

PRIMARY OUTCOMES:
Adverse Event(AE) | From the date of initial infusion to 1 year after initial infusion
  Number of treatment-related adverse events as assessed by CTCAE v4.0
Incidence of bleeding events | From the date of initial infusion to 1 year after initial infusion
  The incidence of bleeding events after initial infusion
The cumulative incidence and grade of graft-versus-host disease (GVHD) including acute and chronic GVHD | From the date of initial infusion to 1 year after initial infusion
  The occurrence incidence and grade of GVHD after transplantation
The probability of GVHD-free, relapse-free survival(GRFS) | From the date of initial infusion to 1 year after initial infusion
  The composite endpoint of GRFS was defined as the first events occurring after transplantation among Grade III to IV aGVHD, moderate to severe cGVHD, relapse, or death for any reason.
Overall response rate (ORR) | 4 weeks after initial infusion
  Percentage of participants achieved Complete response(CR) or Partial response(PR)

SECONDARY OUTCOMES:
Overall response rate (ORR) | 1, 2 and 8 weeks after initial infusion
  Percentage of participants achieved Complete Response(CR) or Partial Response(PR)
Complete remission (CR) rate | 1, 2, 4 and 8 weeks after initial infusion
  CR was defined as a platelet count ≥ 50×10^9/L without platelet transfusions for 7 consecutive days
partial response rate (PR) | 1, 2, 4 and 8 weeks after initial infusion
  PR was defined as a platelet count < 50×10^9/L but above the baseline level at enrollment, with a sustained increase for 7 consecutive days without platelet transfusions
Changes in platelet counts | before treatment and at 1, 2, 4, and 8 weeks after treatment
  Changes in platelet counts before treatment and at 1, 2, 4, and 8 weeks after treatment
Median time of platelet count ≥ 50×10^9/L | 1 year after initial infusion
  Platelet count ≥50×10^9/L for 3 consecutive days without platelet transfusions for 7 consecutive days
Median time of platelet count ≥ 100×10^9/L | 1 year after initial infusion
  Platelet count ≥50×10^9/L for 3 consecutive days without platelet transfusions for 7 consecutive days
Total platelet transfusion during 4 weeks of treatment | 4 weeks after initial infusion
  Total platelet transfusion during 4 weeks of treatment
neutrophil reconstitution | 1 year after initial infusion
  Neutrophil engraftment time was defined as the first of three consecutive days during which the neutrophil count was at least 0.5×10^9/L
erythroid reconstitution | 1 year after initial infusion
  Red blood count (RBC) engraftment time was defined as the first day of achieving a reticulocyte count greater than 1% for 3 consecutive days.
Megakaryocyte levels in bone marrow smears | before treatment and 2 and 4 weeks after treatment
  Megakaryocyte levels in bone marrow smears

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Zhu, Ph.D, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, Anhui, China